CLINICAL TRIAL: NCT02814240
Title: Hepatic Steatosis and Pituitary Gland Failure, Evaluation by NMR Imaging
Brief Title: Hepatic Steatosis and Pituitary Gland Failure, Evaluation by Nuclear Magnetic Resonance (NMR) Imaging
Acronym: SHAH
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire Dijon (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: PETIT NOVARTIS 2014
Record Dates: First submitted 2016-06-23; First posted 2016-06-27 (Estimated); Last update posted 2024-02-21 (Actual); Status verified 2024-02

CONDITIONS: Hepatic Steatosis; Pituitary Gland Failure
MeSH Terms: conditions — Fatty Liver | interventions — Blood Specimen Collection

ARMS (1):
- Pituitary gland failure (Experimental)
  Interventions: Other: NMR; Biological: Blood samples; Other: fibroscan

INTERVENTIONS:
Other: NMR
Biological: Blood samples
Other: fibroscan

SUMMARY:
The investigator put forward the hypothesis that liver fat mass in patients with pituitary gland failure is greater than that in a control population. Failure of the anterior pituitary and more particularly impaired production of growth hormone (GH) could be the principal mechanism responsible for increased liver fat mass in these patients.

ELIGIBILITY:
Inclusion Criteria:

* Patients who have provided consent
* Patients over 18 years
* Patients with pituitary disease (Pituitary adenoma, anterior pituitary failure, craniopharyngioma, empty sella syndrome, hypophysitis, infiltration of the stalk) requiring Magnetic Resonance Imaging (MRI) of the pituitary.

Exclusion Criteria:

* Persons without national health insurance
* Pacemaker (Contra-Indication for MRI)
* Alcohol consumption greater than 4 glasses a day
* Any treatment able to increase liver fat content (glitazones, systemic corticoids, immunosuppressants) are forbidden
* Presence of metallic implants (Contra-Indication for MRI)
* Claustrophobia
* Adult under guardianship
* Pregnant or breast-feeding women
* Patients with a liver disease other than non-alcoholic steatosis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2015-03-16 (Actual); Primary Completion 2015-10-10 (Actual); Study Completion 2015-10-10 (Actual)

PRIMARY OUTCOMES:
Measurement of liver fat mass by Magnetic Resonance Imaging (MRI) | Measured at Day 0

CONTACTS AND LOCATIONS:
Locations (1):
- CHU Dijon Bourgogne, Dijon, France